CLINICAL TRIAL: NCT01254747
Title: Clinical Evaluation of an Investigational Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-347-C-003v2s2v2
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Delefilcon A (Experimental): Delefilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for four weeks.
  Interventions: Device: Delefilcon A contact lens
- Lotrafilcon B (Active Comparator): Lotrafilcon B contact lenses worn in both eyes on a daily wear, daily disposable basis for four weeks.
  Interventions: Device: Lotrafilcon B contact lens (O2 OPTIX, AIR OPTIX)
- Nelfilcon A (Active Comparator): Nelfilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for four weeks.
  Interventions: Device: Nelfilcon A contact lens (DAILIES AquaComfort Plus)
- Narafilcon A (Active Comparator): Narafilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for four weeks.
  Interventions: Device: Narafilcon A contact lens (1-DAY ACUVUE TRUEYE)

INTERVENTIONS:
Device: Delefilcon A contact lens — Investigational silicone hydrogel, single vision contact lens for daily wear, daily disposable use
  Other Names: DAILIES TOTAL1®
  Arms: Delefilcon A
Device: Lotrafilcon B contact lens (O2 OPTIX, AIR OPTIX) — Commercially marketed silicone hydrogel, single vision contact lens for daily wear, daily disposable use
  Other Names: O2 OPTIX®; AIR OPTIX®
  Arms: Lotrafilcon B
Device: Nelfilcon A contact lens (DAILIES AquaComfort Plus) — Commercially marketed hydrogel, single vision contact lens for daily wear, daily disposable use
  Other Names: DAILIES® AquaComfort Plus®
  Arms: Nelfilcon A
Device: Narafilcon A contact lens (1-DAY ACUVUE TRUEYE) — Commercially marketed (Europe) silicone hydrogel, single vision contact lens for daily wear, daily disposable use
  Other Names: 1-DAY ACUVUE® TRUEYE™
  Arms: Narafilcon A

SUMMARY:
The purpose of this 4-week dispensing trial is to evaluate and compare an investigational soft contact lens worn on a daily disposable basis with three other soft contact lenses also worn on a daily disposable basis.

ELIGIBILITY:
Inclusion Criteria:

* Germany: Be of legal age.
* USA: Be of legal age or, if under legal age, have written consent of parent/guardian to participate and sign informed assent.
* Sign Informed Consent.
* Wear soft contact lenses for at least 3 months prior to the study.
* Wear soft contact lenses on a daily disposable basis, daily wear basis, or occasional extended wear basis.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Regularly wear contact lenses on an extended/overnight basis.
* Germany: pregnant or lactating.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- CIBA VISION Research Clinic, Duluth, Georgia, United States
- CIBA VISION Research Clinic, Großwallstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 1 US study center and 1 German study center.
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants (129). One US participant was enrolled, but not dispensed.
Period: Overall Study
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Started | 40 | 29 | 30 | 30
Completed | 40 | 23 | 26 | 28
Not Completed | 0 | 6 | 4 | 2
Not completed — Unacceptable subjective vision | 0 | 0 | 0 | 2
Not completed — Difficult removal handling | 0 | 0 | 1 | 0
Not completed — Symptoms and problems | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Biomicroscopy | 0 | 0 | 1 | 0
Not completed — Discomfort | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A | Total
Number analyzed (Participants) | 40 | 29 | 30 | 30 | 129
Age Continuous [Mean (Standard Deviation); unit: years] — All enrolled and dispensed participants
  years | 35.7 (10.4) | 35.6 (11.4) | 38.4 (10.6) | 37.0 (11.4) | 36.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 19 | 24 | 20 | 95
  Male | 8 | 10 | 6 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall comfort was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: Analysis conducted per protocol, with exclusions due to reasons such as protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Units on a scale | 9.5 (0.7) | 7.9 (1.6) | 9.0 (0.9) | 8.6 (1.2)

2. Primary Outcome: Vision Quality During the Day
Description: Vision quality during the day was assessed and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Vision quality during the day was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Units on a scale | 9.6 (0.6) | 8.8 (1.2) | 9.5 (0.9) | 8.7 (1.3)

3. Primary Outcome: Overall Handling
Description: Overall handling was assessed and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall handling was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Units on a scale | 9.3 (0.9) | 8.5 (1.4) | 9.3 (0.9) | 9.1 (1.3)

4. Primary Outcome: Dryness Throughout the Day
Description: Dryness throughout the day was assessed and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Dryness throughout the day was measured on a 10-point scale, with 1 being very dry and 10 being not dry.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Units on a scale | 9.5 (0.6) | 7.7 (2.0) | 9.0 (1.5) | 8.5 (1.5)

5. Primary Outcome: Average Daily Wear Time
Description: Average daily wear time (hours) was reported by the participant as a single, retrospective evaluation of 4 weeks of wear.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Hours | 13.8 (2.2) | 13.8 (2.1) | 14.2 (1.8) | 13.8 (1.6)

6. Secondary Outcome: Lens Fit
Description: Lens fit was assessed by the investigator for each eye using a biomicroscope, which magnifies the appearance of the contact lens on the participant's eye. Lens fit was graded on a 5-point scale, with 2=unacceptable loose, 1=acceptable loose, 0=optimal, -1=acceptable tight, and -2=unacceptable tight.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Number analyzed (Eyes) | 80 | 46 | 52 | 56
Units on a scale | 0.1 (0.3) | 0.1 (0.6) | 0.1 (0.6) | -0.6 (0.7)

7. Secondary Outcome: Corrected Visual Acuity
Description: Corrected visual acuity was tested for each eye while the participant read distant charts in normal lighting. Corrected visual acuity was measured with a Snellen chart, which was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equates to a logMAR acuity of 0.0 and is considered normal distance eyesight. Positive logMAR values indicate poorer vision, and negative values denote better visual acuity.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Number analyzed (Eyes) | 80 | 46 | 52 | 56
logMAR | -0.06 (0.04) | -0.04 (0.06) | -0.07 (0.05) | -0.06 (0.06)

8. Secondary Outcome: Overall Satisfaction
Description: Overall satisfaction was recorded on a 5-point Likert scale as a single, retrospective evaluation of 4 weeks of wear. The following scale was used: 2=very satisfied, 1=somewhat satisfied, 0=neither, -1=somewhat dissatisfied, and -2=very dissatisfied.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 40 | 23 | 26 | 28
Units on a scale | 1.4 (1.3) | 0.6 (1.4) | 1.5 (0.8) | 1.1 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial: 15-NOV-2010 to 20-DEC-2010.
Description: The safety population included all enrolled and exposed participants: 129.
Arm/Group | Delefilcon A | Lotrafilcon B | Nelfilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/40 | 5/29 | 2/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delefilcon A (N=40) | Lotrafilcon B (N=29) | Nelfilcon A (N=30) | Narafilcon A (N=30)
Contact Lens-Related Discomfort (Eye disorders) | 0 | 5 | 0 | 0
Contact Lens-Related Dryness (Eye disorders) | 0 | 0 | 2 | 0
Contact Lens-Related Unacceptable Subjective Vision (Eye disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes